CLINICAL TRIAL: NCT03774667
Title: Characteristics, Complications and Perinatal Outcomes in Placenta Previa Women: a Prospective, Matched Case-control Study
Brief Title: Characteristics, Complications and Perinatal Outcomes in Placenta Previa Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maternal and Child Health Hospital of Foshan (Other)
Responsible Party: Sponsor
Other Study IDs: MCHHFoshan-1901
Record Dates: First submitted 2018-12-05; First posted 2018-12-13 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Placenta Previa
Keywords: Placenta Previa; Risk Factors; Perinatal Complications; Perinatal Outcomes
MeSH Terms: conditions — Placenta Previa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Placenta Previa: Pregnant women is diagnosed with placenta previa after delivery. Placenta previa is diagnosed by experienced ultrasonologists based on a transabdominal ultrasonic finding of placental tissue covering the internal cervical os before delivery, and further confirmed by obstetricians at delivery.
- None-Placenta Previa: Pregnant women is diagnosed without placenta previa after delivery. Placenta previa is diagnosed by experienced ultrasonologists based on a transabdominal ultrasonic finding of placental tissue covering the internal cervical os before delivery, and further confirmed by obstetricians at delivery.

SUMMARY:
This study aim to investigate the characteristics, complications and perinatal outcomes in pregnant women with placenta previa.

DETAILED DESCRIPTION:
Placenta previa (PP) is defined as the placenta overlying the endocervical os and grades according to the relationship and the distance between the lower placental edge and the internal os of the uterine cervix: low-lying previa, marginal previa, partial previa, and complete previa.

Cesarean delivery and assisted reproductive technology are associated with an increased risk of placenta previa in subsequent pregnancies. Other risk factors for previa include previous spontaneous, elective pregnancy terminations, previous uterine surgery, increasing maternal age and maternal parity, multiple gestations, smoking, cocaine use, and prior previa.

It is associated with numerous adverse maternal and fetal-neonatal complications, such as perinatal hemorrhage, preterm birth, blood transfusion, hysterectomy, maternal intensive care unit admission, disseminated intravascular coagulation, septicemia, thrombophlebitis, and even fetal-neonatal and maternal death.

This is a 1:2 prospective, matched and hospital-based case-control study to investigate the characteristics, complications and perinatal outcomes in pregnant women with placenta previa. For each placenta previa women, the investigators selected two none-placenta previa pregnant women as control from the same department matched on the mode of delivery, using simple random selection when excess matches are available. The date of their admission is limited to two days.

This hospital is a tertiary university-affiliated medical center with a stable number of approximately 12,000 deliveries per year. Placenta previa is diagnosed by experienced ultrasonologists based on a transabdominal ultrasonic finding of placental tissue covering the internal cervical os before delivery, and further confirmed by obstetricians at delivery.

ELIGIBILITY:
Inclusion Criteria:

* Single Pregnancy
* Informed consent
* Fetal gestational age 28 to < 42 weeks

Exclusion Criteria:

* Multiple pregnancy
* Refuses to consent

Ages: 12 Years to 60 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Pregnant women is diagnosed with placenta previa after delivery and their matched pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with postpartum hemorrhage | 24 hours after delivery
  Blood loss > 1000ml during cesarean section or > 500 ml during vaginal delivery

SECONDARY OUTCOMES:
Number of Participants with antepartum hemorrhage | From the time of viability of pregnancy to the delivery of the baby, assessed up to 42 weeks
  At least one episode of bleeding from the genital tract during the antenatal period
Number of Participants with preterm birth | From the time of viability of pregnancy to the delivery of the baby, assessed up to 37 weeks
  Before 37 completed gestational weeks
Number of Participants with very preterm birth | From the time of viability of pregnancy to the delivery of the baby, assessed up to 32 weeks
  Before 32 completed gestational weeks
Number of participant needed for blood transfusion | 72 hours after delivery
  Calculation of the number of participant needed for blood transfusion
Number of urological injury | 72 hours after delivery
  Calculation of the number of participant with bladder or ureteric injury
Number of needed for extra surgical maneuvers | 72 hours after delivery
  internal iliac ligation or hysterectomy
Number of need for caesarean hysterectomy | 72 hours after delivery
  Yes or no
Number of needed for neonatal ICU | 72 hours after delivery
  Yes or no
Number of needed for maternal ICU | 72 hours after delivery
  Yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal and Child Health Hospital of Foshan, Foshan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after completion of the study